CLINICAL TRIAL: NCT06459674
Title: Mean ReSponse Time: Effects of Inspiratory Muscle Training in Postmenopausal Women (MRS)
Brief Title: Inspiratory Muscle Training in Postmenopausal Women
Acronym: MRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Stephen J. Carter, Ph.D., Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20387
Record Dates: First submitted 2024-05-21; First posted 2024-06-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Postmenopausal Symptoms; Aging; Obesity
Keywords: postmenopausal; aging; women's health; blood pressure; mean response time; Inspiratory Muscle Training (IMT)
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All members of the research staff (i.e., those collecting data during experimental visits) will be blinded to the treatment group. The PI, who will not be part of data collection, will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Inspiratory Muscle Training (IMT) group (Experimental): The test protocol requires participants to inhale maximally (maximum inspiratory pressure, MIP) against 2mm diameter leak and sustain inhalation (sustained maximal inspiratory pressure, SMIP) until task failure. Participants will complete 3 SMIP maneuvers with each training session and use the best of the three for that day's training template (corresponding to about 80% SMIP for the IMT group) via the PrO2Fit software. Participants must match or exceed the SMIP template with each increasing level of the work-rest ratio. Work at each level consists of 6 breaths, 36 breaths total. If six breaths are completed, the next level starts. Rest intervals will progressively shorten as training continues from 40-seconds to 5-seconds. The session will be terminated if participants are unable to match at least 90% of the training template for two consecutive breaths or have completed all 36 breaths. Training will be done 4 times a week, and over 8-weeks.
  Interventions: Device: PrO2 Fit (IMT Trainer)
- Sham Inspiratory Muscle Training (Sham-IMT) group (Sham Comparator): Similar to the IMT group protocol, participants will be required to complete 3 SMIP maneuvers with each training session. Participants will use the best of the three for that day's training template (corresponding to about 30% SMIP for the Sham-IMT group) via the PrO2Fit software. Participants must match or exceed the SMIP template with each increasing level of the work-rest ratio. Work at each level consists of 6 breaths, 36 breaths total. If six breaths are completed, the next level starts. Rest intervals will progressively shorten as training continues from 40-seconds to 30-, 20-, 15-, 10-, and 5-seconds. The training session will be terminated if participants are unable to match at least 90% of the training template for two consecutive breaths or have completed all 36 breaths. Training will be done 4 times a week, and over 8-weeks.
  Interventions: Device: PrO2 Fit (IMT Trainer)

INTERVENTIONS:
Device: PrO2 Fit (IMT Trainer) — The device is used four times a week over a period of 8 weeks.

SUMMARY:
This study is being conducted by the Department of Kinesiology within the School of Public Health at Indiana University Bloomington. The purpose of this study is to better understand how inspiratory muscle strength training affects cardiovascular health and mood disturbance in postmenopausal women.

DETAILED DESCRIPTION:
Inspiratory muscle training (IMT) works by strengthening the respiratory muscles through resistive airflow breathing using a handheld device. The goal being to elicit an adaptive response akin to resistance exercise for locomotor muscles. Labored breathing due to respiratory muscle weakness can detract from physical performance with attendant consequences on independent living. This may trigger a maladaptive cycle that worsens physiological and psychosocial outcomes. IMT from 6-10 weeks has been shown to increase maximal inspiratory pressure, functional capacity, and perceived breathlessness across disease states. To inform an appropriately powered randomized controlled trial, the present work proposes a 2-arm single-blind, randomized pilot study to evaluate outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (self-report at least 6 years since last menstrual cycle)
* Aged 50-75 years (confirmed by birth date listed on participant's driver license at screening visit)
* English-speaking
* Body mass index between 25.0 to 39.9 kg/m2
* Able to ambulate without assistance
* Own or have access to a Bluetooth-capable phone or tablet (IOS version 12.0 or later or Android version 7.0 or later)

Exclusion Criteria:

* Unable to provide informed consent.
* Greater than stage II hypertension (i.e., >159/99 mm Hg)
* Current tobacco use (self-report)
* Habitually exercise training ≥ 2 days per week (self-report)
* Significant orthopedic limitations or other contraindications to strenuous exercise
* Live or work > 80 miles from Bloomington, Indiana
* Anticipated elective surgery during the study period.
* Surgery to the chest or abdomen in the last 6 months.
* Plan to move residence or travel out of the local area during the study period.
* History of heart attack or heart condition.
* Current use of prescription medications that affect heart rate or blood vessel dilation (e.g., systemic b-adrenergic blockers, calcium channel blockers, and hormone replacement therapy).
* Diagnosis of asthma or chronic pulmonary disease.
* Current respiratory infection.
* Diagnosis of an aneurysm in the chest, abdomen, or brain.
* Psychological or social characteristics that would interfere with their ability to fully participate in the study.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Duration | Baseline, within 48 hours of completing intervention
  Duration, reported in seconds, to reach 63% of steady-state V̇O2 during a fixed-workload treadmill task. This technique is performed using breath-by-breath open-circuit spirometry and captures the V̇O2 fast component occurring in the transition from standing rest to treadmill walking.

SECONDARY OUTCOMES:
Distance Traveled | Baseline, within 9 days of completing intervention
  Distance traveled, reported in meters, during a 6-minute walk test. The assessment offers reliable and valid insight concerning exercise capacity in older women.

OTHER OUTCOMES:
Cerebral Vascular Reactivity | Baseline, within 9 days of completing intervention
  Cerebral vascular function will be measured in vivo evidenced by changes in cerebral blood flow velocity [i.e., reactivity (cm/s/mm Hg)] of the middle cerebral artery in response to randomized hypercapnic gas exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Carter, Ph.D, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No IDP sharing plan